CLINICAL TRIAL: NCT05261178
Title: Evaluation of Satisfaction With the Use of Myoelectric Controlled Prosthesis and Its Effect on Daily Living Activities in Patients With Upper Extremity Amputation
Brief Title: Evaluation of Satisfaction and Effect on Daily Living Activities With the Use of Myoelectric Controlled Prosthesis
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Gaziler Physical Medicine and Rehabilitation Education and Research Hospital (Other)
Responsible Party: Principal Investigator, Yasin Demir, Physical Medicine and Rehabilitation Specialist, Gaziler Physical Medicine and Rehabilitation Education and Research Hospital
Other Study IDs: 27
Record Dates: First submitted 2022-02-19; First posted 2022-03-02 (Actual); Last update posted 2022-09-30 (Actual); Status verified 2022-02

CONDITIONS: Amputation
Keywords: myoelectric controlled protheses; satisfaction; daily living activities
MeSH Terms: conditions — Personal Satisfaction

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Upper extremity amputation patients using myoelectric controlled prosthesis: 20 patients aged 18-65 years with upper extremity amputation and using myoelectric controlled arm prosthesis for at least 3 months
  Interventions: Other: Evaluation of satisfaction and the level of daily living activities using the prosthesis

INTERVENTIONS:
Other: Evaluation of satisfaction and the level of daily living activities using the prosthesis — Evaluation of satisfaction with using the prosthesis with TAPES (Trinity Amputation and Prosthesis Experience Scale) and the level of daily living activities using the prosthesis with SF-36 (Short Form-36)

SUMMARY:
Myoelectrically controlled arm prostheses are often offered to individuals with upper extremity limb loss in order to restore body balance and compensate for the lack of grasping ability during the rehabilitation process. Myoelectrically controlled prostheses utilize the presence of two independent signals from a set of agonist and antagonist muscles. However, individuals with upper extremity amputation may not want to use their prosthesis. One of the reasons for not wanting to use the prosthesis is prosthesis dissatisfaction. This study aims to evaluate prosthesis satisfaction and the effect of prosthesis use on daily living activities of upper extremity amputees using myoelectric controlled prosthesis.

DETAILED DESCRIPTION:
The study will be carried out with patients who applied to the outpatient clinic or who received inpatient treatment in the orthopedic rehabilitation (amputee) clinic. The patient's demographic information (age, gender, height, weight, body mass index, education level, occupation, marital status) and clinical characteristics (amputation date, cause of injury, amputation side, etc.) will be recorded with the evaluation to be made to the patient. Patients' satisfaction with using their prosthesis will be evaluated with TAPES (Trinity Amputation and Prosthesis Experience Scale) and daily living activities using their prosthesis with SF-36 (Short Form-36).

ELIGIBILITY:
Inclusion Criteria:

1. Being between the ages of 18-65
2. Having an upper extremity amputation
3. Using myoelectric controlled arm prosthesis for at least 3 months

Exclusion Criteria:

1. Being under the age of 18
2. Having significant cognitive or hearing impairment that would preclude participation in research

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 20 patients aged 18-65 years with upper extremity amputation and using myoelectric controlled arm prosthesis for at least 3 months
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2022-10-01 (Estimated); Primary Completion 2022-10 (Estimated); Study Completion 2022-10-01 (Estimated)

PRIMARY OUTCOMES:
Trinity Amputation and Prosthesis Experience Scale | Through study completion, an average of one and a half months
  It consists of two parts after the first part, which includes demographic and disability-related information. Part I covers psychosocial adjustment, activity restriction, and satisfaction with the prosthesis. In the second part, there are questions about how many hours a day the prosthesis is worn on average, general health status and physical capacity. The scores are summed up with a subscale score between 10 and 50. Higher scores correspond to satisfaction with the prothesis.
SF-36 (Short Form-36) | Through study completion, an average of one and a half months
  It consists of eight scales (general health, physical function, physical role, emotional role, social function, pain, energy, mental health), each varying between 2-10 questions, and a health course question that is not included in the scoring. Each question is scored on only one scale. Scoring is made between 0-100 for each scale. The lowest score represents the worst health condition.

CONTACTS AND LOCATIONS:
Overall Officials: Fatma Özcan, MD, Principal Investigator — Gaziler Physical Medicine and Rehabilitation Education and Research Hospital